CLINICAL TRIAL: NCT04448730
Title: Can the Betatrophin be a Reliable Marker of Insulin Resistance in Normal Weight and Overweight Women With Polycystic Ovary Syndrome?
Brief Title: Polycystic Ovary Syndrome and BETATROPHIN
Status: Completed | Type: Observational
Sponsor: Hatice Akkaya (Other Government)
Responsible Party: Sponsor-Investigator, Hatice Akkaya, associate professor, Kayseri Education and Research Hospital
Organization: Kayseri Education and Research Hospital (Other Government)
Other Study IDs: EZTB24
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2019-01

CONDITIONS: Polycystic Ovary; Obesity
Keywords: Betatrophin; PCOS; obesity; insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (normal weight with PCOS ): 35 cases
  Interventions: Diagnostic Test: serum marker levels
- overweight PCOS: 38 cases
  Interventions: Diagnostic Test: serum marker levels

INTERVENTIONS:
Diagnostic Test: serum marker levels — two groups comparisons

SUMMARY:
This is an original study giving an information about the association body mass index, polycystic ovary syndrome and betatrophin.

DETAILED DESCRIPTION:
Introduction: Betatrophin is a protein hormone which has a significant role in glucose homeostasis and lipid metabolism. The aim of this study is to compare the levels of serum betatrophin in overweight and normal weight women with PCOS.

Material and Method: Thirty-five patients normal weight women with PCOS (BMI<25) and 38 obese women with PCOS (BMI≥25) were included in this prospective, cross-sectional study. Patients were selected according to Rotterdam criteria. Serum betatrophin levels were studied by ELISA method and then compared between these two groups besides the following additional parameters as waist circumference/hip circumference ratio, fasting blood glucose, 75 g OGTT (oral glucose tolerance test) results and HOMA-IR levels.

ELIGIBILITY:
Inclusion Criteria:

-Polycystic ovary syndrome according to 2003 Rotterdam PCOS Consensus diagnostic criteria

Exclusion criteria

* pregnancy,
* an additional systemic disease (i.e.,hyperprolactinemia, thyroid dysfunction, liver or kidney diseases, cardiovascular disease, hyperlipidemia, type 1 or type 2 diabetes, chronic or acute infection within the previous 30 days),
* morbid obesity,
* smoking,
* the use of medications for contraception, androgen excess, hypertension, hyperglycemia or dyslipidemia at least 3 months before the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Comparison of the Betatrohin serum marker of insulin resistance in normal weight and overweight women with polycystic ovary syndrome cases.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
serum Betatrophin levels | 30 min
  ng/L

SECONDARY OUTCOMES:
Waist/hip ratio | 5 min
  centimeter
75 gr OGTT(oral glucose tolerance test) | 2 hours
  (mg/dl)
BMI (body mass index) | 5 minute
  kg/m2

CONTACTS AND LOCATIONS:
Locations (1):
- Kayseri Doğumevi, Kocasinan, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
If needed
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: journals editors request